CLINICAL TRIAL: NCT07290829
Title: Conformity of Conjunctival Hyperemia Assessment in Soft Contact Lens Wearers Using Image J Analysis and Efron Degree System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Tri Rahayu, SpM(K), FIACLE, MD, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-02-0138; Faculty of Medicine, Universit (Other: Faculty of Medicine, Universitas Indonesia)
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Soft Contact Lenses
Keywords: soft contact lens; conjunctival hyperemia; image J analysis; efron degree system

STUDY DESIGN:
Masking Description: Conjunctival inflammation degree evaluation was done with taking picture of conjunctiva using slit lamp by lead researcher. Picture was taken on day 0 (before using SCL), day 7, and day 14 of wearing SCL. Pictures then were analyzed with Efron Degree System (EDS) by 2 evaluators (both were ophthalmologist consultants) and with ImageJ application by lead researcher. ImageJ analysis was done to decide conjunctival vascular diameter and density. EDS evaluator did not know the results of the assessment with ImageJ and vice versa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Hyperemia evaluation of soft contact lens wearer (Experimental): Hyperemia evaluation of soft contact lens wearer on day 0 (before using SCL), day 7, and day 14 of wearing SCL
  Interventions: Device: hydrogel soft contact lens

INTERVENTIONS:
Device: hydrogel soft contact lens — This study aim to analyze the conformity of hyperemia when evaluated by ophthalmologist using the Efron degree system compared to evaluation by a computerized model (Image J analysis )

SUMMARY:
Soft Contact Lens (SCL) use all over the world is still increasing. Ocular surface inflammatory reaction is the most common risk of using SCL. Currently, the standard used to assess this complication is the Efron Degree System (EDS), but it has high variability due its subjectivity. ImageJ gives more objective result with conjunctival vasodilation and vascular density assessment, so that complication management can be given earlier.

Purpose: Evaluate the suitability of SDE with ImageJ analysis in assessing conjunctival hyperemia in SCL use within 2 weeks.

DETAILED DESCRIPTION:
This is a paired prospective analytic study. Subjects with myopia who have not used SCL routinely before were instructed to use SCL for 14 days. Conjunctival inflammation were assessed with slit lamp examination before, at day 7, and day 14 of using SCL. Slit lamp pictures were analysed with EDS and ImageJ to be compared.

ELIGIBILITY:
Inclusion Criteria:

* subject with mild to moderate myopia (-0.50 to -6.00 D)
* age between 18-45 years old
* subject who refuse refractive correction with glasses or surgery
* patient with astigmatism refractive error no more than -1 Diopter

Exclusion Criteria:

* subject with previous intraocular surgery
* subject who is wearing SCL continuously
* subject with history of dry eyes, uveitis, glaucoma, or corneal and conjunctival disorders
* subject with history of allergic reaction to contact lens material or lens wetting solution used in this study
* subject with ongoing eye drop treatment
* female subject with ongoing pregnancy or on breastfeeding
* subject with too improper lens fitting
* subject who work around exposure of chemical substance, smoke, hazardous gas, or fire sparks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Efron degree system for hyperemia degree | on day 0 (before using SCL), day 7, and day 14
  Hyperemia grade based on Efron degree system, identified by percentage of hyperemia on the bulbar dan limbal conjunctiva
  * Normal
  * Trace
  * Mild
  * Moderate
  * Severe
Image J analysis of hyperemia degree | on day 0 (before using SCL), day 7, and day 14
  Vascular density (%area) and Vascular diameter (μm )

CONTACTS AND LOCATIONS:
Overall Officials: Tri Rahayu, MD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital
Locations (1):
- Department of Ophthalmology, Faculty of Medicine Universitas Indonesia Cipto Mangunkusumo Hospital, Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient privacy considerations